CLINICAL TRIAL: NCT06425952
Title: Impact of Sensory, Motor and Vestibular Deficit on the Postural Stability of CMT Patients
Acronym: EquiCMT
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Stefano Previtali, Head Neuromuscular Repair Unit, IRCCS San Raffaele
Other Study IDs: OSRSCP-EquiCMT
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Hereditary Neuropathy
Keywords: CMT neuropathy; equilibrium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CMT patients: patients with sensory-motor genetic neuropathy
- Motor patients: Patients with motor genetic neuropathy
- Sensory patients: Patients with sensory neuropathy
- Myopathic patients: Patients with distal myopathy

SUMMARY:
Charcot-Marie-Tooth (CMT), a therapeutically orphan neuromuscular disease affecting one in 2,500 people, represents a challenge to the medical and scientific communities. Physiotherapeutic-rehabilitative strategies play a crucial role in the management of CMT, particularly addressing balance impairment, a key disabling symptom. However, clinical studies in this field are limited. Our study aims to investigate the impact of strengh and somatosensory deficits on static and dynamic balance in CMT patients. The Investigators also aim to explore the involvement of the vestibular system and its correlation with postural instability. Furthermore, the Investigators seek to evaluate relationships between neurochemical biomarkers offering valuable insights for future targeted clinical studies.

DETAILED DESCRIPTION:
A total of 60 patients will be recruited. To ensure adequate representation of the subgroups of interest, 10 patients with CMT1A (PMP22 gene duplication) and 10 patients with CMT2, regardless of their genotype, will be included. Additionally, three control groups, each comprising 10 subjects, will be included. The first group will consist of patients with motor symptoms, including those with hereditary motor neuropathy (HMN, 10 patients) or distal myopathy (MD, 10 patients). The second group will include patients with solely sensory symptoms, genetic neuropathies, or purely sensory acquired neuropathies such as HSN and neuropathies from anti-MAG antibodies. Finally, the third group will be composed of 10 healthy subjects. Each control subject will have comparable level of disability (motor or somatosensory), age, and gender to the enrolled CMT patients.

All participants must meet the following inclusion criteria to take part in the study:

* Age 18 years or older
* Subject has documented diagnosis of one of the following diseases (except from healthy controls):

  * Hereditary sensory-motor neuropathy (CMT) confirmed by genetic analysis
  * Hereditary motor neuropathy (HMN) confirmed by genetic analysis
  * Hereditary sensory neuropathy (HSN) confirmed by genetic analysis
  * Hereditary distal myopathy (MD) confirmed by genetic analysis
  * Acquired sensory neuropathy: anti-MAG antibody neuropathy confirmed by neurophysiological, clinical and serological assessment.

The presence of any one of the following exclusion criteria will lead to the exclusion of the subject:

* Inability to maintain an upright position without assistance
* Presence of systemic, neurological (except for the neuropathies and hereditary myopathies under study), psychiatric, orthopedic or rheumatological diseases that may affect evaluation
* Mini Mental State Examination (MMSE)14 score less than 28
* History of alcohol or substance abuse
* Partecipation in intensive motor rehabilitation programs in the last three months.

ELIGIBILITY:
Inclusion Criteria:

* CMT or HMN or sensory neuropathy or distal myopathy

Exclusion Criteria:

* unable to stand
* other neurological, psychiatric, or orthopedic disorders
* MMSE <28
* alcohol abuse
* intensive rehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 CMT1A patient, 10 CMT2, 10 HMN, 10 sensory neuropathies, 10 distal myopathies, 10 healthy controls.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Postural equilibrium | 12 months
  How sensory and motor deficit influence the postural equilibrium

SECONDARY OUTCOMES:
Vestibular equilibrium | 12 months
  how vestibular system influence the postural equilibrium

CONTACTS AND LOCATIONS:
Overall Officials: Stefano C Previtali, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- Dept. of Neurology, IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No